CLINICAL TRIAL: NCT04803253
Title: Evaluating the Relevance of Social and Professional Reintegration Improvements With a Set of Solutions for People With Upper Limb Amputation: Longitudinal Analysis of 2 Cohorts in Selected Areas of Nepal.
Brief Title: Study of the Social and Professional Reintegration Improvements Using a Set of Solutions for Upper Limb Amputation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orthopus (Industry)
Collaborators: Handicap International (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CST-0404-201006
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Amputation; Traumatic, Arm, Upper; Amputation; Traumatic, Arm: Forearm; Amputation; Traumatic, Hand, at Wrist Level; Wounds and Injuries
Keywords: amputation; transradial; prosthesis; terminal device; upper limb amputation; upper extremity
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants using the ORTHOPUS set of prosthetic solution (Experimental)
  Interventions: Device: ORTHOPUS prosthetic accessory: 0109 - Universal Wrist; Device: ORTHOPUS prosthetic terminal device: 0112 - Hook; Device: ORTHOPUS prosthetic terminal device: 0105 - Cosmetic Articulated Hand; Device: ORTHOPUS prosthetic accessory: 0104 - body powered harness

INTERVENTIONS:
Device: ORTHOPUS prosthetic accessory: 0109 - Universal Wrist — The ORTHOPUS mechanical wrist device is intended to provide an external wrist joint only for external upper limb prostheses with pronation/supination passive motion (activation with external force), a quick connection (with automatic lock) and manual disconnection of the mechanical wrist connectors.
  The mechanical wrist connector allows to quickly switch between different type of terminal devices (hand or tools).
Device: ORTHOPUS prosthetic terminal device: 0112 - Hook — The ORTHOPUS body-powered hook is a Voluntary Opening (VO) device made of aluminium intended to provide high grasping capabilities under harsh environments.
Device: ORTHOPUS prosthetic terminal device: 0105 - Cosmetic Articulated Hand — The ORTHOPUS cosmetic articulated hand is intended to provide a replacement limb in order to hide the loss of the original one. It is composed of an aesthetic glove (18 colors and 3 sizes, silicone made) and of an internal structure that can be bent to achieve a given position allowing the user to grasp small and light objects.
Device: ORTHOPUS prosthetic accessory: 0104 - body powered harness — The ORTHOPUS body powered harness is intended to allow the patient to actuate the 0112 - Hook device. It will be installed on the patient's contralateral shoulder and linked to the 0112 - Hook device with a cable.

SUMMARY:
ORTHOPUS develops assistive technologies to address the lack of availability of medical devices in low and middle income countries.

With the help of HI (Handicap International) Nepal, the need for upper limb prostheses was identified. Indeed, according to the literature - especially Efficiency of voluntary opening hand and hook prosthetic devices: 24 years of development? (JRRD, Volume 49, Number 4, 2012) -, today available solutions do not fully address patients' needs.

In Nepal, only 2 upper limb prostheses options are generally proposed to patients because of supply and cost constraints.

ORTHOPUS' objective is to extend patients' autonomy with a new set of prosthetic solutions. By offering low cost but high quality devices (according to CE marking requirements), another of the ORTHOPUS' missions is also to address supply and cost constraints.

To improve patients' capabilities, ORTHOPUS aims at extending grasping capabilities compared to the usual passive aesthetic hand or voluntary opening one by proposing the following set of solutions:

* an aesthetic articulated hand
* a mechanical wrist
* a work hook

In order to assess the different stated hypotheses, a clinical trial is set jointly with HI Nepal. 14 patients will be enrolled in 2 cohorts (n1 = 7, n2 = 7), the first one is constituted with patients usually using an aesthetic passive hand whereas the second one comprise patients normally equipped with voluntary opening hand.

After selecting and getting the informed consent of the patients, a month to make the sockets and adapt it to patients is planned. An evaluation of their quality of life will be done with the WHO QOL - BREF quality of life assessment before and after the test period of the trial.

ORTHOPUS' set of prosthetic solutions will be tested by them over one month. They will have to fill on a daily basis a survey (OPUS) assessing their use of the prostheses. At the end of the test period, different questionnaires and surveys will be filled during a last interview to collect data.

Data will be analysed in order to extract evidence for or against the trial hypotheses. With these results, a report will be written and submitted to the GATE (Global Cooperation on Assistive Health Technology) community managed by WHO. This report will also feed the ORTHOPUS R&D with patients' feedbacks and, research findings will be shared publicly on different social media in respect with patient privacy.

DETAILED DESCRIPTION:
BACKGROUND

ORTHOPUS is a french private company founded in 2018 with the mission of increasing access to assistive technology like prosthetics care. ORTHOPUS focuses its actions on low and middle income countries with a model that mixes social impact (open source, frugal innovation, fair pricing) and medical european quality (CE marking).

Today, over 1 billion people need at least one form of Assistive Technology (AT), but over 900 million people (90%) do not have access to the AT they require.

The number of people who need AT is expected to grow to more than 2 billion people by 2050 according to the WHO "Assistive Technology Fact Sheet 18 May 2018". 80% of these persons live in a Low or Middle Income Country (LMIC).

According to World Health Organization estimation, 0.5% of the populations need these services and a report from the United Nations highlights that 0.7% of the Nepalese populations are physically disabled - NEPAL: Disabled Population 2011, (UNRCHCO, 2011). Prosthetics and Orthotics (P&O) service is the subset of rehabilitation service, and National health policy 2019 has identified rehabilitation as core health services .

Compared to other assistive products such as crutches and walkers, P&O services are very scarcely available in Nepal, even-though its need is going higher due to the increasing prevalence of NCDs and road traffic injury.

Living Conditions among People with Disability in Nepal report (SINTEF, 2015) highlights that 73 percent of people with disabilities do not have access to Assistive Devices.

According to WHO, failure of health policies, excessive prices of products, provision difficulties and insufficient training of health personnel are the 4 reasons for this problem.

RATIONALE

ORTHOPUS objective is to address some of the problem highlighted by WHO:

* To address LMIC product-related problems, ORTHOPUS proposes quality prosthetic solutions with a moderate price by designing innovative solutions based on the frugal innovation concept
* To address Information transmission and Health care practitioner formation, all ORTHOPUS' solutions will be shared via a free/Open source licence
* In order to guarantee the quality of medical devices, ORTHOPUS follows European standards certification process for each and every product.

Nepal is one of the target countries of the ORTHOPUS objective as the 2011 Nepal Census conducted by the government of Nepal reported that 1.94% of the total population of Nepal is living with some kind of disabilities. The number will be more if the 'functioning' status of the population is considered.

Moreover, the Living Conditions among People with Disability in Nepal report (SINTEF, 2015) highlights that 83 percent of people with disabilities do not have access to rehabilitation services and that there is a 72.5% service gap in Assistive Devices.

Today, according to the Principal Investigator of the trial, the most popular solutions provided by healthcare practitioners, in LMICs such as Nepal, for transradial amputation is a voluntary opening hand or a passive aesthetics one.

The voluntary opening hand is a compromise between efficiency and aesthetics according to the publication Efficiency of voluntary opening hand and hook prosthetic devices: 24 years of development? (JRRD, Volume 49, Number 4, 2012).

On the other hand, the passive aesthetic solution does not provide any active grasping functionalities but has an important social impact for users hiding the limb loss to a certain extent.

In addition, Nepal was chosen for ORTHOPUS first clinical trial thanks to the help of HI (Humanity and Inclusion) NGO who has already a program there. HI staff, Yeti Raj Niraula, will be the principal investigator of this clinical trial.

This clinical trial will focus on upper-limb prostheses. ORTHOPUS wants to demonstrate that a set of solutions composed of multiple medical devices such as:

* a wrist with a possible pronosupination as well as a rotational lock and a quick connection/disconnection feature.
* an aesthetic articulated hand, similar to usual aesthetic passive hand proposed nowadays in Nepal but with an additional articulation feature
* a heavy duty work hook used as a working tool to address the shortage of heavy duty prosthetic products in the country. The trial aims at assessing if using this solution will improve work integration of the user.
* a harness used to actuate the work hook allowing the user to open it with muscular contraction of the upper part of the torso

With this trial, improvement of the autonomy of users and on the well-being in everyday life will be studied compared to the sole use of a voluntary opening hand or a passive aesthetics one.

GENERAL OBJECTIVE

The general objective is to show the relevance of using the set of solutions made by ORTHOPUS (aesthetic articulated hand, working hook and quick disconnect wrist) compared to the widespread solution of a voluntary opening hand or passive aesthetic one.

SPECIFIC OBJECTIVE

To establish the effect of the ORTHOPUS prosthetic solution, four primary objectives will be studied to address the scientific question by collecting appropriate data:

* improvement of grasping capacities
* improvement of quality of life
* improvement of sociodemographic conditions
* evaluation of prosthesis perception

To address the primary objectives of the trial the following subjective primary endpoints will be measured:

* improvement of grasping capacities will be evaluated using an adapted to Nepali culture OPUS survey (Development and measurement properties of the Orthotics and Prosthetics Users' Survey (OPUS): a comprehensive set of clinical outcome instruments, A W Heinemann, 2003). Participants will be ranking the ease of realisation of a 30 item list using ORTHOPUS prosthetic solution. These ranks will be compared to the one obtained using the previous prosthetic solution (if applicable). Studying results to the survey, a conclusion on the evolution of the grasping capacities of users will be formulated.
* improvement of quality of life will be evaluated using the WHOQoL-BREF questionnaire (World Health Organisation, Program of Mental Health. WHOQOL-BREF : introduction, administration, scoring and generic version of the assessment : field trial version. 1996). Participants will be asked to answer 27 questions with ranked propositions before and after the test phase of the clinical trial. Scores will be compared to evaluate improvements brought by the ORTHOPUS prosthetic solution on the quality of life of the user and a conclusion will be drawn.
* improvement of sociodemographic conditions will be evaluated using a questionnaire written following the guidance of guidelines Standardization and Harmonization of Socio-Demographic Variables (2016, GESIS Survey Guidelines). Again a comparison of the answers to the 28 entries of the form will be made confronting questionnaires filled before and after the clinical trial test phase.
* evaluation of prosthesis perception will be conducted using a questionnaire filled by participants at the end of the test phase of the clinical trial. Analysis of the ranks given to the 90 entries will allow to draw a precise picture of the participants' perception of the ORTHOPUS prosthesis solution. With these results a conclusion will be drawn on the ORTHOPUS' solution improvements that needs to be performed to improve future users' perception.

Results of evaluations of objectives achievements will be used to feed ORTHOPUS' R&D department in order to improve the studied prosthetic solution or to launch development of new products.

RESEARCH HYPOTHESIS

Nowadays, in Nepal, most of the patients are equipped with either a voluntary opening hand or a passive aesthetic one. These solutions present grasping capabilities or aesthetics limitations (see additional document attached to the registration: Comparative scheme - Standard VS ORTHOPUS prosthetic solutions.pdf) and we hypothesize that the ORTHOPUS prosthetic solution will expand it.

In addition with this grasping capabilities expansion, we hypothesize that, compared to previously used prosthetic solution, the set of ORTHOPUS upper limb prosthetics solutions will:

* improve the autonomy of users (professional reintegration with the ability to perform manual work)
* improve the well-being in everyday life (social reintegration)

For the patient selection, we hypothesize that two different cohorts will be enough to discriminate the data and make good clinical trial conclusions.

The first cohort will be composed of prosthetic users usually equipped with aesthetic passive hand solutions. The second one with a voluntary opening hand user. Data gathered from both cohorts will allow a direct comparison between the use of voluntary opening hand or passive aesthetic one (according to the cohort) and the use of the ORTHOPUS prosthetic solution.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transradial or wrist-disarticulation amputee
* 20 to 50 years of age
* At least 1 year from date of amputation
* Have been using upper limb prosthesis previously
* Be able to independently provide informed and independant consent
* Be willing to comply with study procedures
* Independent function by self-report
* Free of any health ailment that would impair physical function

Exclusion Criteria:

* Congenital anomaly of upper limb
* Bilateral wrist disarticulation or transradial amputation
* Any condition that would prevent participation and pose increased risk (e.g. shoulder impingement, sub-acromial bursitis, severe arthritis of the shoulder, elbow, wrist, or fingers)
* Injuries of the upper limb within the past 90 days (surgeries, sprains, strains, or fractures).
* Younger than 20 or older than 50 years of age
* Unwillingness/inability to follow instructions
* History of acute or chronic skin breakdown on the residual limb
* Any health ailment that would impair physical function

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Functionalities of the prosthetic solution | 1 month
  Users' feedback will be gathered from his/her experiences and quantitative data will be collected using the "OPUS Upper Extremity Functional Status" survey, which allows us to evaluate the contribution of the set of solutions to the accomplishment of daily life tasks. For each activity, the user will evaluate the difficulty of performing the activity (very easy; easy; slightly difficult; very difficult; cannot perform the task; not applicable), and will specify whether or not he or she usually uses his or her prosthesis in performing the task.
Quality of life evolution | 1.5 month
  Quality of life will be evaluated with the "WHO QOL - BREF quality of life assessment". The form is composed of checkboxes entries ranking from: very low, low, neither good nor low, good, very good. Users will have to fill in the form twice: once before the patient testing and a then at the end of it. This will allow a comparison of the results and the determination of a potential improvement.
Prosthesis perception | 1.5 month
  Prosthesis perception will be evaluated with a final questionnaire created by ORTHOPUS to collect users' feedback on aesthetics, functionalities and sensations. These aspects will be evaluated with scores from 1 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: David Gouaillier, PhD, Study Director — Orthopus
Locations (3):
- Nepal (3):
  - Prerana Rehabilitation Center, Sarlahi, Malangawa
  - Community Based Rehabilitation, Biratnagar
  - Social Welfare Council - National Disabled Fund, Kathmandu

IPD SHARING:
Plan to Share IPD: No